CLINICAL TRIAL: NCT04619680
Title: Early Nintedanib Deployment in COVID-19 Interstitial Lung Disease
Brief Title: The Study of the Use of Nintedanib in Slowing Lung Disease in Patients With Fibrotic or Non-Fibrotic Interstitial Lung Disease Related to COVID-19
Acronym: ENDCOV-I
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Maria L Padilla, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 20-2147
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Fibrosis; Interstitial Lung Disease; Respiratory Disease
Keywords: COVID-19; Infiltrates; SARS CoV-2; lung; scarring; fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Respiration Disorders; COVID-19; Cicatrix; Fibrosis | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: * Patients will be assigned to nintedanib or placebo by random chance in a 1:1 allocation. There is 50% chance to receive the study drug and a 50% chance to receive the placebo.
  * Randomization will be stratified by site and subgroup (fibrotic and non-fibrotic) to ensure treatment balance. I.e., within the fibrotic subgroup, the randomization will ensure 50% are assigned to the nintedanib arm and 50% are assigned to the placebo arm. Similarly, treatment balance within the non-fibrotic subgroup will be ensured.
  * The study will be double blinded. No one (including the patient or the study team) will know who is receiving the study drug or the placebo. If it becomes urgently necessary for a patient's care, the study doctor will be able to find out whether the patient is taking the placebo or the study drug, nintedanib.
  * Patients will be told whether they received the study drug, nintedanib, or the placebo once the study is finished.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nintedanib (Experimental): 150 mg PO twice a day, taken with food, (or, for Child-Pugh A patients, 100 mg by mouth twice daily).
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): placebo equivalent 150mg PO twice a day, taken with food food (or, for Child-Pugh A patients, 100 mg by mouth twice daily).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — 150 mg PO twice a day, taken with food food (or, for Child-Pugh A patients, 100 mg by mouth twice daily).
  Arms: Nintedanib
Drug: Placebo — placebo 150 mg equivalent twice a day, taken with food food (or, for Child-Pugh A patients, 100 mg by mouth twice daily).
  Arms: Placebo

SUMMARY:
This is a collaborative study between Icahn School of Medicine at Mount Sinai, Boehringer Ingelheim Pharmaceuticals and up to 9 other clinical centers across the US to determine the effect of nintedanib on slowing the rate of lung disease in patients who have been diagnosed with COVID-19, and have ongoing lung injury more than 30 days out from their diagnosis. Required one of the following after diagnosis with SARS-CoV-2: supplemental oxygen by nasal cannula, high flow oxygen, non invasive ventilation such as CPAP or BIPAP, or mechanical ventilation or a history of desaturation below 90%.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of the study drug, nintedanib, on slowing the rate of lung disease in patients who are noted to have infiltrates, or ongoing lung injury, on chest x-ray/CT 30 days or longer from their initial symptoms. In addition, the study will also investigate patient reported outcomes using questionnaires, and the safety and tolerability of the study drug. Blood specimens will be collected to assess biomarkers and monitor drug safety.

The trial will be randomized 1:1 between nintedanib and placebo.

Nintedanib has been approved by the FDA for the treatment of chronic fibrosing ILD with a progressive phenotype, but has not been studied in patients with post COVID 19 lung disease.

Subjects participating in this study will:

* Attend in person visits to the study doctor's office on the date of enrollment, 15 days after enrollment, 45 days after enrollment, 90 days after enrollment, 135 days after enrollment, and 180 days after enrollment. If the participant is being enrolled in the study while hospitalized, the study doctor will travel to the hospital room. There will also be a follow-up phone call 30 days after finishing study drug.
* Undergo a HRCT (High-resolution computed tomography) scan of the chest within 6 weeks of enrollment, and then again at 180 days after enrollment.
* Have Pulmonary Function Tests within 14 days of enrollment, and then again 45, 90, 135 and 180 days after enrollment.
* Have a six-minute walk test at baseline, day 90 and day 180 after enrollment.
* Have blood drawn routinely while participating in this study (within 14 days of randomization, 15 days after starting medication, then again on day 45, 90, 135 and 180).
* Participants will not pay for physician visits, blood draws, breathing tests, CT scans or the medication for this study. Participants will receive a stipend to cover the transportation costs for your visits.

The main risks to participants are:

1. Common side effects include: nausea, vomiting, diarrhea, stomach discomfort
2. Loss of appetite and weight loss
3. Liver function abnormalities (blood work will be monitored periodic intervals at scheduled blood draws as listed above)
4. Slightly higher risk of bleeding
5. Slightly higher risk of blood clots that can form in the blood vessels that supply oxygen to vital organs such as the brain and heart
6. Kidney disease resulting in protein/and or albumin being lost through urine

Benefits from participation in this research include the possibility that nintedanib may slow down/prevent progression of lung fibrosis. If the lungs can heal without fibrosis, this may result in fewer symptoms of shortness of breath, cough and need for added oxygen.

Instead of participating in this research, subjects may choose to monitor their lung condition with their doctor or participate in another research study.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Subjects Age ≥ 18
* Initial SARS-CoV-2 infection confirmed by PCR test or positive serologies
* Have findings consistent with interstitial lung disease found on CT scan (these may include ground glass opacities, reticulations, traction bronchiectasis, septal thickening, and early honeycombing)
* Required one of the following after diagnosis with SARS-CoV-2: supplemental oxygen by nasal cannula, high flow oxygen, non invasive ventilation such as CPAP or BIPAP, or mechanical ventilation or a history of desaturation below 90%
* Are at least 30 days from onset of initial SARS-CoV-2 symptoms
* Forced Vital Capacity less than or equal to 90% predicted based on ATS/ERS criteria or DLCO less than or equal to 70%
* Women of childbearing potential who agree to use of highly effective contraception during treatment and for three months following the last dose of nintedanib

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of the Screening Visit (prior to randomization):

* Co-administration of other investigational agents against COVID-19
* Active SARS-CoV-2 infection based on clinical judgment
* Currently Pregnant or Breast Feeding
* Current Use of Prednisone or equivalent > 10 mg/daily or immunosuppressive therapy or disease modifying agents
* Use of full dose anticoagulation therapy or high dose anti platelet drug therapy at screening (at the discretion of the investigator, anticoagulation therapy may be added if clinically indicated)
* History of myocardial infarction within past 90 days
* Life threatening bleed
* Hemodynamic instability or shock
* Superimposed pulmonary bacterial infection
* Pre-existing interstitial lung disease
* Active Hep A/B/C hepatitis as measured with PCR for viral load and/or serologies
* Pre-existing liver disease: Including Abnormal Laboratory Liver Function: Childs Pugh B/C, AST/ALT > 3 times the upper limit of normal (ULN). If Child Pugh A, can participate on nintedanib 100 mg by mouth twice daily.
* Subjects with a Creatinine clearance <30 ml/min or currently on hemodialysis
* Inability to tolerate orally administered medication (medication must be taken with meals)
* Patients who are in the intensive care unit (ICU) or in the step-down unit on invasive or non-invasive mechanical ventilation, ECMO, or high flow nasal cannula oxygen, will not be included.
* Any condition that in the opinion of the Investigator, constitute a risk or a contraindication for the participation of the patient into the study or that could interfere with the study objectives, conduct or evaluation.
* Patients with known hypersensitivity to nintedanib, peanut, soy, or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-02 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Baseline and 180 days
  Change in Forced Vital Capacity (FVC) at 180 days as compared to baseline. Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry.

SECONDARY OUTCOMES:
Number of deaths due to respiratory cause | within 90-180 days
  Death within 90 days and 180 days from enrollment due to a respiratory cause
Chest CT visual score | 180 days
  Quantitative Change in chest CT visual score graded by blinded chest radiologists. Data driven texture analysis (DTA) is a patented deep learning method to quantify lung fibrosis. DTA score is reported in percentage ranging from 0% to 100%. A minimally clinical important difference when comparing CT scans from the same subject is 4%. A higher percentage suggests worsening lung injury.
St. George's Respiratory Questionnaire (SGRQ) | Day 90
  The Saint George's Respiratory Questionnaire (SGRQ) is a self-reported disease-specific, health-related quality of life (QOL) questionnaire. 50-item instrument. Scores range from 0 to 100, with higher scores indicating more limitations.
St. George's Respiratory Questionnaire (SGRQ) | Day 180
  The Saint George's Respiratory Questionnaire (SGRQ) is a self-reported disease-specific, health-related quality of life (QOL) questionnaire. 50-item instrument. Scores range from 0 to 100, with higher scores indicating more limitations.
King's Brief Interstitial Lung Disease Questionnaire (KBILD) | Day 90
  The King's Brief Interstitial Lung Disease (KBILD) questionnaire is a self-administered, ILD-specific measure of health-related quality of life, comprising 15 items with three domains (Psychological (KBILD-P), Breathlessness and activities (KBILD-B), and Chest symptoms (KBILD-C)) combined in a total score (KBILD-T). The KBILD domain and total score ranges are 0-100; 100 represents best health status.
King's Brief Interstitial Lung Disease Questionnaire(KBILD) | Day 180
  The King's Brief Interstitial Lung Disease (KBILD) questionnaire is a self-administered, ILD-specific measure of health-related quality of life, comprising 15 items with three domains (Psychological (KBILD-P), Breathlessness and activities (KBILD-B), and Chest symptoms (KBILD-C)) combined in a total score (KBILD-T). The KBILD domain and total score ranges are 0-100; 100 represents best health status.
Leicester Cough Questionnaire (LCQ) | Day 90
  The LCQ is a 19 item questionnaire that assesses cough-related QOL. It has 3 domains (physical, psychological and social). The domain scores range from 1-7 and total score range is 3-21 with a higher score indicating a better quality of life.
Leicester Cough Questionnaire (LCQ) | Day 180
  The LCQ is a 19 item questionnaire that assesses cough-related QOL. It has 3 domains (physical, psychological and social). The domain scores range from 1-7 and total score range is 3-21 with a higher score indicating a better quality of life.
Short Form (SF) 36 Health Survey | Day 90
  The (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status. Scores range from 0 - 100, with higher scores indicating less disability.
Short Form (SF) 36 Health Survey | Day 180
  The (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status. Scores range from 0 - 100, with higher scores indicating less disability.
Hospital Anxiety and Depression Scale (HADS) | Day 90
  Questionnaire with 7 items for anxiety and 7 items for depression, each item is scored on a 4 point response 0 - 3, with full range from 0 to 42, with higher score indicating more severe anxiety or depression.
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Hospital Anxiety and Depression Scale (HADS) | Day 180
  Questionnaire with 7 items for anxiety and 7 items for depression, each item is scored on a 4 point response 0 - 3, with full range from 0 to 42, with higher score indicating more severe anxiety or depression.
  14-items scale with responses scored from 0-3, scores for each subscale from 0 (normal) to 21 (severe symptoms). Scores for the entire scale is 0 to 42, with higher score indicating more distress.
Number of participants with Increase in liver transaminases (AST and ALT) > 3 times the upper limit of normal | day 90
  Number of participants with Increase in liver transaminases
Number of participants with Increase in liver transaminases (AST and ALT) > 3 times the upper limit of normal | day 180
  Number of participants with Increase in liver transaminases
Number of participants with Thrombotic events | day 90
  Number of participants with Thrombotic events: venous or arterial thrombosis
Number of participants with Thrombotic events | day 180
  Number of participants with Thrombotic events: venous or arterial thrombosis
Number of participants with 10% weight loss over 90 days | day 90
  Number of participants with 10% weight loss
Number of participants with 10% weight loss over 90 days | day 180
  Number of participants with 10% weight loss
Number of participants with GI events | day 90
  Number of participants with Nausea/emesis/diarrhea not responsive to anti-emetics and anti-motility agents
Number of participants with GI events | day 180
  Number of participants with Nausea/emesis/diarrhea not responsive to anti-emetics and anti-motility agents
Change in 6 minute walk test | Baseline and day 180
  The distance covered over a time of 6 minutes at day 180 as compared to baseline.
Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) | Day 90
  The FACIT-F is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Questions are scored on a 5-point Likert scale. The total score range is from 0-52, with higher score indicating lower fatigue level.
Functional Assessment of Chronic Illness Therapy- Fatigue (FACIT-F) | Day 180
  The FACIT-F is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. Questions are scored on a 5-point Likert scale. The total score range is from 0-52, with higher score indicating lower fatigue level.
Change in Forced Vital Capacity (FVC) | Baseline and Day 90
  Change in Forced Vital Capacity (FVC) at 90 days as compared to baseline. Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry.
Change in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) | Baseline and Day 180
  Change in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) at 180 days as compared to baseline. Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) measures the transfer of carbon monoxide from alveolar gas to hemoglobin in pulmonary capillary blood. DLCO is measured by having the patient fully inhale a low concentration of carbon monoxide and an inert tracer gas.
Number of deaths due to any cause | within 90-180 days
  Number of deaths within 90 days and 180 days from enrollment due to a any cause

CONTACTS AND LOCATIONS:
Overall Officials: Maria Padilla, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - Emory Healthcare Network, Atlanta, Georgia
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor University Medical Center Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals should be directed to Maria.Padilla@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website

REFERENCES:
- [Derived] Santibanez V, Mathur A, Zatakia J, Ng N, Cohen M, Bagiella E, Brown SA, Rosas IO, Patel NM, Olson A, Li P, Padilla M. Early nintedanib deployment in COVID-19 interstitial lung disease (ENDCOV-I): study protocol of a randomised, double-blind, placebo-controlled trial. BMJ Open Respir Res. 2025 Apr 10;12(1):e002323. doi: 10.1136/bmjresp-2024-002323. PMID 40216412